CLINICAL TRIAL: NCT05036668
Title: An Open Label Cryptosporidium Controlled Human Infection Model (CHIM) to Assess the Efficacy and Safety of ABO809 in Healthy Participants
Brief Title: Study of Efficacy and Safety of ABO809 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CABO809A02101
Record Dates: First submitted 2021-08-31; First posted 2021-09-05 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-06

CONDITIONS: Cryptosporidium Infection, Cryptosporidiosis
Keywords: Controlled Human Infection Model, safety, tolerability, healthy volunteers, cryptosporidiosis, ABO809
MeSH Terms: conditions — Cryptosporidiosis

STUDY DESIGN:
Intervention Model Description: Cryptosporidium controlled human infection model
Masking Description: Open-Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ABO809 (Experimental): Participants will receive ABO809 at a single oral dose of 1x10^4 oocysts. Other doses such as 1x10^6 oocysts may be considered to optimize the model
  Interventions: Biological: Cryptosporidium parvum oocysts (ABO809)

INTERVENTIONS:
Biological: Cryptosporidium parvum oocysts (ABO809) — ABO809 3x10^6 CE/3mL concentrate for oral suspension, single dose at Day 1

SUMMARY:
The purpose of this Phase I controlled human infection model (CHIM) study was to determine if oral administration of a good manufacturing practice (GMP) supply of Cryptosporidium parvum oocysts (ABO809) to healthy volunteers resulted in a Cryptosporidium infection and diarrheal illness. The study measured fecal oocysts (parasitological endpoint) as well as diarrhea and associated signs and symptoms (clinical endpoint).

DETAILED DESCRIPTION:
This study was funded by the Wellcome Trust. This Phase 1 Cryptosporidium controlled human infection model (CHIM) study employed a single-center, open-label design to characterize the incidence of infection and associated symptoms following the administration of single doses of Cryptosporidium parvum oocysts (CE).

Healthy volunteers were enrolled in cohorts of approximately 10 participants who received ABO809 on the same day (Day 1). The study consisted of three sequential cohorts which were dosed one after the other for a total of 30 participants. A dose level group received the same ABO809 dose and could be comprised of multiple cohorts. The first dose level group started with a cohort of 10 participants who received ABO809 at a dose of 1x10^4 oocysts. The study continued to enroll participants in the same dose level group if the desired incidences of infection and diarrheal illness were observed, up to a total of approximately 30 participants. If the desired incidences of infection and diarrheal illness were not observed, a new dose level group, receiving ABO809 at a dose of 1x10^6 oocysts, could be initiated. If needed to optimize the model, intermediate ABO809 doses could be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Demonstrated understanding of Cryptosporidium disease, safety measures and transmission risks
* Good health
* Ability to communicate well with the Investigator

Exclusion Criteria:

- History of Cryptosporidium infection, gastrointestinal conditions (including diarrheal syndromes, gastroenteritis and gastrointestinal tract surgery), immunodeficiency, infections, significant medical concerns, hypersensitivity to nitazoxanide or other specified antibiotics.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-07 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-12-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Al-Ibrahim, Principal Investigator — Pharmaron CPC, Inc.
Locations (1):
- Novartis Investigative Site, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in one investigative site in one country.
Groups:
- ABO809 1x10^4 CE-Cohort 1: ABO809 single oral dose of 1x10^4 oocysts.
- ABO809 1x10^6 CE-Cohort 2; ABO809 1x10^6 CE-Cohort 3: ABO809 single oral dose of 1x10^6 oocysts.
Period: Overall Study
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Started | 10 | 10 | 10
Completed | 10 | 10 | 9
Not Completed | 0 | 0 | 1
Not completed — lost to follow Up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3 | Total
Number analyzed (Participants) | 10 | 10 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (6.53) | 33.4 (7.03) | 34.1 (8.49) | 33.9 (7.15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 2 | 13
  Male | 5 | 4 | 8 | 17
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 6 | 5 | 8 | 19
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 1
  White | 3 | 4 | 1 | 8
  Other | 0 | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Cryptosporidium Infection From 72 Hours to 10 Days Post ABO809 Oral Administration
Description: Cryptosporidium infection was measured by examining the presence of a Cryptosporidium antigen in stool using a commercially available diagnostic Enzyme Immunoassay (EIA) test. Up to 3 stool samples per day were collected, each separated by approximately 4-hour intervals, were analyzed by EIA for parasitological assessment of oocyst shedding.
Time Frame: At ≥72 hours post-administration (or sooner if associated with symptoms suggestive of diarrheal illness) up to Day 10 (inclusive).
Population: The pharmacodynamic (PD) analysis set included all participants with available parasitological and clinical data and with no protocol deviations with relevant impact on PD data.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Number analyzed (Participants) | 10 | 7 | 10
percentage of participants | 50 [26.73 to 73.27] | 57.1 [27.86 to 83.04] | 60.0 [35.42 to 81.24]

2. Secondary Outcome: Percentage of Participants Showing Clinical Diarrheal Illness From Day 1 to Day 28 Post ABO809 Oral Administration
Description: Clinical diarrheal illness was defined as the occurrence of at least two diarrheal bowel events within 24 hours on at least two days after the administration of ABO809. Diarrhea is defined as at least one stool sample grading 3-5 on the Stool Grading system in one day. Grades 1 and 2 are considered normal stool and Grades 3-5 are considered diarrheal stool.
  Grade 1 stool is defined as formed stool which does not take the shape of the container.
  Grade 2 stool is defined as soft stool which does not easily take the shape of the container.
  Grade 3 diarrheal stool is defined as thick liquid stool taking the shape of the container.
  Grade 4 diarrheal stool is defined as opaque watery stool. Grade 5 diarrheal stool is defined as rice water or clear watery stools.
Time Frame: From Day 1 up to Day 28
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Number analyzed (Participants) | 10 | 7 | 10
percentage of participants
  Clinical diarrheal illness up to Day 10 (inclusive) | 60.0 [35.42 to 81.24] | 57.1 [27.86 to 83.04] | 50.0 [26.73 to 73.27]
  Clinical diarrheal illness up to Day 28 (inclusive) | 60.0 [35.42 to 81.24] | 57.1 [27.86 to 83.04] | 50.0 [26.73 to 73.27]

3. Secondary Outcome: Number of Diarrhea Stools Per Participant
Description: Diarrhea is defined as at least one stool sample grading 3-5 on the Stool Grading system in one day. Grades 1 and 2 are considered normal stool and Grades 3-5 are considered diarrheal stool.
  Grade 1 stool is defined as formed stool which does not take the shape of the container.
  Grade 2 stool is defined as soft stool which does not easily take the shape of the container.
  Grade 3 diarrheal stool is defined as thick liquid stool taking the shape of the container.
  Grade 4 diarrheal stool is defined as opaque watery stool. Grade 5 diarrheal stool is defined as rice water or clear watery stools.
Time Frame: From Day 1 up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Error); unit: diarrheal stools
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Number analyzed (Participants) | 10 | 7 | 10
diarrheal stools | 13.3 (4.85) | 16.2 (7.15) | 12.9 (3.41)

4. Secondary Outcome: Overall Diarrheal Stool Weight
Description: Stool weight in grams of each stool from each participant were measured during inpatient period from Day 1 up to Day 10. Stool weight in grams of stool collected 24 hours prior to outpatient visit from each participant were measured during outpatient period from Day 14 to Day 28.
Time Frame: From Day 1 up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Number analyzed (Participants) | 10 | 7 | 10
grams | 1614.0 (1541.84) | 2681.6 (2798.02) | 2877.0 (1884.71)

5. Secondary Outcome: Maximum Stool Grade by Stool Grade Category
Description: All collected stool samples were graded according to the Stool Grading system. Grades 1 and 2 are considered normal stool and Grades 3-5 are considered diarrheal stool. Grades 3-5 stools are defined as thick liquid diarrhea taking the shape of the container, opaque watery, rice water or clear watery stools. The maximum stool grade is the highest stool grade of all episodes in a participant.
Time Frame: From Day 1 up to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Number analyzed (Participants) | 10 | 7 | 10
Participants
  Stool Grade 1 | 0 | 0 | 1
  Stool Grade 2 | 2 | 2 | 3
  Stool Grade 1 and 2 | 2 | 2 | 4
  Stool Grade 3 | 3 | 1 | 1
  Stool Grade 4 | 2 | 1 | 2
  Stool Grade 5 | 3 | 3 | 3
  Stool Grade >= 3 | 8 | 5 | 6

6. Secondary Outcome: Time to Onset of Clinical Diarrheal Illness
Description: Clinical diarrheal illness was defined as the occurrence of at least two diarrheal bowel events within 24 hours on at least two days after the administration of ABO809. The time to onset is the number of days until the start diarrheal illness.
Time Frame: From Day 1 up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Number analyzed (Participants) | 6 | 4 | 5
days | 3.3 (1.97) | 3.3 (0.96) | 2.8 (0.45)

7. Secondary Outcome: Time to Resolution of Clinical Diarrheal Illness
Description: Clinical diarrheal illness was defined as the occurrence of at least two diarrheal bowel events within 24 hours on at least two days after the administration of ABO809. The time to resolution is the number of days until the resolution of diarrheal illness, which is defined as 2 or more consecutive days with no diarrheal stools (stool grades 1 or 2).
Time Frame: From Day 1 up to Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Number analyzed (Participants) | 6 | 4 | 5
days | 9.0 (1.26) | 9.8 (2.22) | 10.0 (3.54)

8. Secondary Outcome: Percentage of Participants With Characteristics of Clinical Signs and Symptoms Associated With Clinical Diarrheal Illness
Description: Clinical signs and symptoms associated with clinical diarrheal illness such as: abdominal pain, abdominal cramping, nausea, vomiting, fever, electrolyte disbalance, dehydration.
Time Frame: From Day 1 up to Day 28
Population: Safety analysis set (SAF) included all participants that received one dose of ABO809 during the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Number analyzed (Participants) | 10 | 10 | 10
Participants
  Abdominal discomfort | 1 | 0 | 0
  Abdominal distension | 3 | 0 | 1
  Abdominal pain | 5 | 7 | 2
  Abdominal tenderness | 0 | 2 | 1
  Defaecation urgency | 4 | 2 | 4
  Flatulence | 1 | 2 | 2
  Haematochezia | 1 | 3 | 2
  Nausea | 3 | 4 | 1
  Rectal tenesmus | 0 | 0 | 1
  Vomiting | 1 | 5 | 1
  Pyrexia | 1 | 2 | 2
  Occult blood | 1 | 1 | 0
  Occult blood positive | 1 | 0 | 1
  Decreased appetite | 2 | 6 | 4
  Dehydration | 2 | 2 | 2

9. Secondary Outcome: Percentage of Participants With Cryptosporidium Infection From 72 Hours to Day 28 Post ABO809 Oral Administration
Description: Percentage of participants with Cryptosporidium infection following an oral administration of ABO809. Cryptosporidium infection were measured by examining the presence of a Cryptosporidium antigen in stool using a commercially available diagnostic Enzyme Immunoassay (EIA) test.
Time Frame: From 72 hours post-administration up to Day 28
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Number analyzed (Participants) | 10 | 7 | 10
percentage of participants | 60.0 [35.42 to 81.24] | 57.1 [27.86 to 83.04] | 60 [35.42 to 81.24]

10. Secondary Outcome: Percentage of Participants With Fecal Shedding of Cryptosporidium Parvum Oocysts
Description: Percentage of participants with fecal shedding of Cryptosporidium parvum oocysts following an oral administration of ABO809. Fecal shedding will be measured by examining the presence of a Cryptosporidium antigen in stool using a commercially available diagnostic Enzyme Immunoassay (EIA) test.
Time Frame: From 72 hours post-administration up to Day 28
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: percentage of participants
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Number analyzed (Participants) | 10 | 7 | 10
percentage of participants | 60.0 [35.42 to 81.24] | 57.1 [27.86 to 83.04] | 60.0 [35.42 to 81.24]

11. Secondary Outcome: Time to Onset of Cryptosporidium Infection
Description: Time to onset is the number of days until the start of Cryptosporidium infection which were measured by examining the presence of a Cryptosporidium antigen in stool using a commercially available diagnostic Enzyme Immunoassay (EIA) test.
Time Frame: From Day 1 up to Day 10
Population: The pharmacodynamic (PD) analysis set included all participants with available parasitological and clinical data and with no protocol deviations with relevant impact on PD data. Only participants with an actual infection were included in the analysis.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Number analyzed (Participants) | 5 | 4 | 6
days | 4.0 (0.71) | 4.0 (0.0) | 4.0 (0.0)

12. Secondary Outcome: Time to Resolution of Cryptosporidium Infection
Description: Time to resolution is the number of days until the resolution of Cryptosporidium infection in participants who developed an infection following an oral administration of ABO809. Resolution of Cryptosporidium infection is defined as no evidence of Cryptosporidium in stool samples collected over ≥2 consecutive days.
Time Frame: From Day 1 up to Day 28
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: days
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Number analyzed (Participants) | 5 | 4 | 6
days | 10.6 (2.61) | 10.8 (2.50) | 9.7 (1.86)

13. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESIs)
Description: The following adverse events associated with Cryptosporidium infection are considered AESIs in this trial: Gastroenteritis in the absence of Cryptosporidium infection, extraintestinal cryptosporidiosis, persistent or recurrent cryptosporidiosis, persistent cryptosporidium shedding, moderate or severe dehydration and non-intestinal sequelae including eye pain or joint pain.
Time Frame: Adverse events were reported from oral administration of ABO809 up to a maximum duration of 56 days.
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | ABO809 1x10^4 CE-Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3
Number analyzed (Participants) | 10 | 7 | 10
Participants
  Participants with AESI | 2 | 2 | 2
  Moderate or severe dehydration | 2 | 2 | 2
  Gastroenteritis in the absence of Cryptosporidium infection | 0 | 0 | 0
  Extraintestinal cryptosporidiosis | 0 | 0 | 0
  Persistent or recurrent cryptosporidosis | 0 | 0 | 0
  Persistent cryptosporidium shedding | 0 | 0 | 0
  Non-intestinal sequelae including eye pain or joint pain | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from oral administration of ABO809 up to a maximum duration of 56 days.
Groups:
- ABO809 1x10^4 CE - Cohort 1: ABO809 single oral dose of 1x10^4 oocysts.
- ABO809 1x10^6 CE - Cohorts 2 and 3: ABO809 single oral dose of 1x10^6 oocysts.
- Total: Total
Arm/Group | ABO809 1x10^4 CE - Cohort 1 | ABO809 1x10^6 CE-Cohort 2 | ABO809 1x10^6 CE-Cohort 3 | ABO809 1x10^6 CE - Cohorts 2 and 3 | Total
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/20 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 0/10 | 0/20 | 0/30
Other Adverse Events (participants affected / at risk) | 10/10 | 9/10 | 9/10 | 18/20 | 28/30
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ABO809 1x10^4 CE - Cohort 1 (N=10) | ABO809 1x10^6 CE-Cohort 2 (N=10) | ABO809 1x10^6 CE-Cohort 3 (N=10) | ABO809 1x10^6 CE - Cohorts 2 and 3 (N=20) | Total (N=30)
Palpitations (Cardiac disorders) | 1 | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 6 | 3 | 9 | 9
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 3 | 0 | 1 | 1 | 4
Abdominal pain (Gastrointestinal disorders) | 6 | 7 | 2 | 9 | 15
Abdominal tenderness (Gastrointestinal disorders) | 0 | 2 | 1 | 3 | 3
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 2 | 3
Defaecation urgency (Gastrointestinal disorders) | 4 | 2 | 4 | 6 | 10
Diarrhoea (Gastrointestinal disorders) | 8 | 8 | 6 | 14 | 22
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 2
Flatulence (Gastrointestinal disorders) | 2 | 2 | 2 | 4 | 6
Haematochezia (Gastrointestinal disorders) | 1 | 3 | 3 | 6 | 7
Nausea (Gastrointestinal disorders) | 3 | 4 | 1 | 5 | 8
Proctalgia (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 1
Rectal tenesmus (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 5 | 1 | 6 | 7
Chills (General disorders) | 1 | 0 | 2 | 2 | 3
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 1
Pain (General disorders) | 2 | 1 | 0 | 1 | 3
Pyrexia (General disorders) | 1 | 2 | 2 | 4 | 5
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 1 | 1 | 2
Body temperature increased (Investigations) | 0 | 3 | 0 | 3 | 3
Heart rate increased (Investigations) | 1 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 1 | 1 | 1
Occult blood (Investigations) | 1 | 1 | 0 | 1 | 2
Occult blood positive (Investigations) | 1 | 0 | 1 | 1 | 2
Decreased appetite (Metabolism and nutrition disorders) | 2 | 6 | 4 | 10 | 12
Dehydration (Metabolism and nutrition disorders) | 2 | 2 | 2 | 4 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 4 | 7
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 2 | 2 | 4 | 4
Headache (Nervous system disorders) | 5 | 6 | 4 | 10 | 15
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 1
Hot flush (Vascular disorders) | 0 | 0 | 1 | 1 | 1
Hypotension (Vascular disorders) | 0 | 1 | 0 | 1 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT05036668/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT05036668/SAP_001.pdf